# Low-Level Laser in Treatment of Head and Neck Lymphedema: A Pilot Study

Principal Investigator Jie Deng, PhD, RN, OCN, FAAN

Department of Biobehavioral Health Sciences University of Pennsylvania School of Nursing

215-573-2393

jiedeng@nursing.upenn.edu

**Co-Investigator** Alexander Lin, MD

**Department of Radiation Oncology** 

The Hospital of the University of Pennsylvania

215-662-3198

Co-Investigator/Statistician Alexandra Hanlon, PhD

Department of Biobehavioral Health Sciences University of Pennsylvania School of Nursing

215-898-4581

Co-Investigator John Nicholas Lukens, MD

Assistant Professor of Radiation Oncology

Department of Radiation Oncology

The Hospital of the University of Pennsylvania

# **Table of Contents**

# **Contents**

| LI | ST OF ABBREVIATIONS | IV |
|---|---|---|
| S | TUDY SUMMARY | 1 |
| В | ACKGROUND AND STUDY RATIONALE | 2 |
| | 1 INTRODUCTION | 3<br>3<br>3 |
| 2 | STUDY OBJECTIVES | 3 |
| | 2.1 PRIMARY OBJECTIVE | 3 |
| 3 | INVESTIGATIONAL PLAN | |
| | 3.1 GENERAL DESIGN 3.1.1 Screening Phase 3.1.2 Study Intervention Phase and Follow Up Phase 3.2 STUDY ENDPOINTS. 3.2.1 Primary Study Endpoints 3.2.2 Secondary Study Endpoints | 4<br>4<br>4 |
| 4 | STUDY POPULATION AND DURATION OF PARTICIPATION | 4 |
| | 4.1 INCLUSION CRITERIA 4.2 EXCLUSION CRITERIA 4.3 SUBJECT RECRUITMENT 4.4 DURATION OF STUDY PARTICIPATION 4.5 TOTAL NUMBER OF SUBJECTS AND SITES 4.6 VULNERABLE POPULATIONS | 4<br>4<br>5 |
| 5 | STUDY INTERVENTION (STUDY DRUG, DEVICE, BIOLOGIC, VACCINE, FOOD ETC.) | 5 |
| | 5.1 DESCRIPTION. 5.2 INTERVENTION REGIMEN 5.3 STORAGE. 5.4 PREPARATION AND PACKAGING 5.5 BLINDING. 5.6 SUBJECT COMPLIANCE MONITORING. | 5<br>5<br>5 |
| 6 | STUDY PROCEDURES AND DATA COLLECTION | 6 |
| | 6.1 SCREENING 6.2 STUDY INTERVENTION PHASE 6.2.1 Visit 1: Baseline Visit 6.2.2 Visit 2: End of Intervention 6.2.3 Visit 3: 4 – Week post Intervention 6.3 SUBJECT WITHDRAWAL | 6<br>6<br>6 |
| 7 | STATISTICAL PLAN AND STATISTICAL ANALYSIS | 7 |
| 8 | SAFETY AND ADVERSE EVENTS | 7 |
| | 8.2 RECORDING OF ADVERSE EVENTS | 7 |

| Version | n: 06-15-2019 | 9 |
|---|---|---|
| | REPORTING OF ADVERSE EVENTS, ADVERSE DEVICE EFFECTS AND UNANTICIPATED PROBLEM | IS TO PENN |
| IRB | 3 AND ACC | 8 |
| | 8.3.1 Investigator reporting: notifying the study sponsor | |
| | STOPPING RULES | |
| | MEDICAL MONITORING | |
| ٥ | 8.5.1 Data and Safety Monitoring Plan | 8 |
| 9 5 | STUDY ADMINISTRATION, DATA HANDLING AND RECORD KEEPING | 9 |
| 9.1 | CONFIDENTIALITY | 9 |
| 9.2 | | |
| 10 5 | STUDY MONITORING, AUDITING, AND INSPECTING | 9 |
| 10. | 1 STUDY MONITORING PLAN | 9 |
| 10.2 | | |
| 11 E | ETHICAL CONSIDERATIONS | 10 |
| 11. | 1 Risks | 10 |
| 11.3 | 2 Benefits | 10 |
| 11.3 | | |
| 11.4 | 4 INFORMED CONSENT PROCESS / HIPAA AUTHORIZATION | 11 |
| 12 5 | STUDY FINANCES | 11 |
| 12. | 1 Funding Source | 11 |
| 12.2 | | |
| 12.3 | 3 SUBJECT PAYMENTS | 11 |
| 13 E | BENCHMARKS FOR STUDY/PUBLICATION PLANPLAN | 11 |

# **List of Abbreviations**

**CDT:** Complete decongestive therapy

HNC: Head and neck cancer

**LLLT:** Low-level laser therapy

**Study Summary** 

| Study Summary | |
|---|---|
| Title | Low-Level Laser in Treatment of Head and Neck Lymphedema: A Pilot Study |
| Short Title | Low-level laser therapy in head and neck lymphedema |
| Study ID Number | UPCC12318 |
| Protocol Number | Version Date: 06-15-2019 |
| Phase | Pilot study |
| Methodology | A single-arm, pre- and post-design clinical trial |
| Study Duration | 24 months |
| Study Center(s) | Single-center |
| Objectives | Primary aim: To determine the feasibility of the use of LLLT for HNC survivors with lymphedema, specifically to 1) obtain recruitment estimates and determine barriers to recruitment; 2) identify barriers to implementation; 3) assess safety; and 4) evaluate patient satisfaction. Secondary aim: To determine the preliminary efficacy of the use of LLLT on the following outcomes: 1) lymphedema progression; 2) symptom burden; and 3) functional status. |
| Number of Subjects | 25 subjects expected to be enrolled |
| Main Inclusion and<br>Exclusion Criteria | Inclusion criteria: >18 years of age; 2) completion of either postoperative radiation or chemoradiation therapy; 3) no evidence of cancer; 4) having head and neck external lymphedema; 5) ability to speak and read English; and 6) able to provide informed consent. Patients will be excluded if they have any of the following medical conditions that would prohibit the safe implementation of LLLT: pregnancy; photosensitivity; chronic inflammatory diseases; venous thrombosis; history of severe trauma; medication that affects body fluid and electrolyte balance; use of high doses of non-steroidal anti-inflammatory drugs; or pre-existing skin rash, ulceration, open wound in the treatment area; and allergic and other systemic skin diseases. |
| Investigational device For Device include the planned use | RianCorp LTU-904 Low-level laser therapy unit |
| Duration of administration (if applicable) | 6 weeks |
| Safety Evaluations | Common Terminology Criteria for Adverse Events (CTCAE version 4.03) will be used to document adverse events of the clinical trial |
| Data and Safety<br>Monitoring Plan | PI Deng will be responsible for monitoring the data quality and the ongoing safety of subjects. |

### **BACKGROUND AND STUDY RATIONALE**

This study will be conducted in full accordance all applicable University of Pennsylvania Research Policies and Procedures and all applicable Federal and state laws and regulations including the use of a medical device (i.e., RianCorp LTU-904).

### 1 Introduction

Current standard of care for head and neck lymphedema treatment provided by therapists is short-term in nature (usually up to 4-12 weeks); however, lymphedema is a chronic condition and often worsens over time. Therefore, alternative treatment modalities need to be investigated for effective and long-term management of lymphedema and associated late fibrosis in the head and neck cancer (HNC) population.

# 1.1 Background and Relevant Literature

There has been an increase in the incidence of head and neck cancer (HNC) largely related to the epidemic of human papillomavirus (HPV) associated disease. 1.2 HPV- associated HNC occurs in younger and middle-aged patients; cure rates in this population are markedly higher compared to other HNC groups. 3.4 This contributes to more than half a million HNC survivors in the U.S. today. 5 Regardless of cause, patients with locally advanced HNC are usually treated with aggressive multi-modality regimens.6 These regimens often lead to numerous long-term toxicities. One common but under-treated late effect of treatment is damage to lymphatic structures and soft tissues resulting in lymphedema. 7.8 Animal studies indicate that lymphedema is associated with chronic inflammation leading to fibrosis. 9,10 Our work was the first to assess lymphedema in HNC patients in a systematic manner. 7,11 We demonstrated a prevalence rate of 75% in HNC survivors. We confirmed that lymphedema occurs both externally (e.g., face and neck) and internally (e.g., pharynx and larynx).7,12 Subsequent work demonstrated that external lymphedema resulted in a decreased range of motion in the jaw, neck and shoulders. 13 Internal swelling was found to cause substantial impact on critical functions (e.g., swallowing, speaking, and breathing). 13,14 Psychological effects (e.g., body image disturbance) were also correlated with lymphedema. 13,15-17 Finally, lymphedema has the potential to negatively impact HNC survivors' ability to function in both home and work environments, resulting in both emotional and financial burden for these individuals, their families, and the healthcare system. 11,18

Current standard of care for treatment of lymphedema is complete decongestive therapy (CDT), which consists of 4 main parts: manual lymphatic drainage, compression (bandaging or garments), exercise, and skin care. <sup>10,19,21,22</sup> These treatments are expensive, time-consuming and labor-intensive. CDT provided by therapists is short-term in nature (usually up to 4-12 weeks); however, lymphedema is a chronic condition and often worsens over time. <sup>10,19</sup> Therefore, alternative treatment modalities need to be investigated for effective and long-term management of lymphedema and associated late fibrosis in the HNC population.

Among many alternative treatment options, low level laser therapy (LLLT) is a promising, noninvasive modality for treatment of lymphedema. LLLT, also named photobiomodulation therapy (PBMT), has had a place in general medicine for more than 40 years.<sup>24</sup> It has been used as a treatment option to stimulate wound healing and reduce inflammation, edema, and pain.<sup>24</sup> The U.S. Food and Drug Administration (FDA) accepted it as a treatment approach for breast cancer-related upper extremity lymphedema (BCRL) in 2006.<sup>24</sup> One recent systematic review evaluating 7 randomized clinical trials (RCT) concluded that available evidence supports LLLT in the management of BCRL, with clinically meaningful reductions in lymphedema-related swelling and symptom burden (e.g., pain).<sup>25</sup> Compared to other treatment modalities, LLLT is a noninvasive modality, repeatable, easily performed in outpatient setting, and without any known long-term side effects. To our knowledge, the current proposal is the first study investigating the use of LLLT in the treatment of head and neck lymphedema. The goal of this proposed research is to determine the feasibility and preliminary efficacy of the use of LLLT on facial/neck swelling and fibrotic changes, symptom burden, and neck mobility in HNC survivors with lymphedema through a pilot study.

### Name and Description of the Investigational Product

We will use a RianCorp LTU-904, FDA-approved, Class I laser device in this study. The device will be used by the study lymphedema therapist, Joy Cohen, who has had more than 20 years of experience treating individuals with lymphedema.

### 1.2.1 Nonclinical Data

Findings from nonclinical data indicate that LLLT stimulates lymphatic vessels and lymphocytes, as well as increases local fluid circulation.<sup>27,28</sup>

### 1.2.2 Clinical Data to Date

Currently, only cases studies indicate the potential value of use of LLLT for treating head and neck lymphedema.<sup>29,30</sup> No large prospective clinical trials are available to evaluate prophylactic and/or therapeutic use of LLLT for lymphedema in HNC patients. However, a large body of evidence is available in supporting the safety and efficacy of LLLT for management of lymphedema in breast cancer patients. For instance, since 1995, the use of LLLT has been investigated in the treatment of breast cancer-related lymphedema (BCRL).31 A meta-analysis of 9 studies (7 of them were RCTs) provided evidence that LLLT alone or combined with other treatments was able to reduce the arm swelling and pain in women with BCRL.31 LLLT does not increase the risk on cellulitis, a known side effect in patients with arm lymphedema.31 A recent systematic review also suggested the use of LLLT for treating the following conditions in the breast cancer population: oral mucositis, radiodermatitis, chemotherapy-induced peripheral neuropathy, and osteonecrosis of the jaw.<sup>24</sup> In another recent systematic review, the authors concluded that LLLT may have potential applications in the management of a broad range of side effects (e.g., lymphedema/fibrosis) of chemo-radiation therapy in patients with HNC.32,33

### 1.2.3 Clinical Studies in Children

Not applicable

### 1.3 Dose Rationale (if applicable)

We propose that participants will receive LLLT twice a week for 6 weeks (12 sessions). This regimen was developed based on the evidence from literature.

### 2 **Study Objectives**

The goal of this proposed research is to evaluate the effect of LLLT on facial/neck swelling and fibrotic changes, symptom burden, and neck mobility in HNC survivors with lymphedema through a pilot study.

### 2.1 **Primary Objective**

To determine the feasibility of the use of LLLT for HNC survivors with lymphedema.

#### 2.2 Secondary Objective

To determine the preliminary efficacy of the use of LLLT for HNC survivors with lymphedema.

### 3 **Investigational Plan**

## General Design

We will conduct a single-arm, pre-and post-design clinical trial. Outcome measures include: 1) feasibility (barriers to implementation, safety, and satisfaction) of the proposed intervention [Primary aim]; and 2) preliminary efficacy (lymphedema progression, symptom burden, and functional status) of the proposed intervention [Secondary aim]. Study assessments will take place at baseline, immediately after end of the intervention, and 4-week post-intervention.

### 3.1.1 Screening Phase

We will recruit a minimum of 6 participants per month. The volume of HNC patients at Penn's Clinic is sufficient to complete this trial without additional sites. The following recruitment procedures will be used: screening at HNC clinics and attendance at Head and Neck tumor board and case conferences. All direct patient recruitment activities will be conducted at the Penn HNC clinics where private rooms are available to be used for conducting clinical research projects.

### 3.1.2 Study Intervention Phase and Follow Up Phase

After completion of the baseline measures, participants will be scheduled for LLLT. The LLLT includes receiving LLLT twice a week for 6 weeks (12 sessions) (LLLT protocol developed based on the literature review<sup>34-41</sup>). After completion of the 12-session LLLT, participants will be given a) contact information and instructions to call for problems and b) a calendar outlining dates for 4-week follow-up data collection.

### 3.2 Study Endpoints

# 3.2.1 Primary Study Endpoints

The primary endpoint will be the feasibility of LLLT in HNC patients, including recruitment estimates, barriers to recruitment, and barriers to implementation, safety, as well as patient satisfaction.

# 3.2.2 Secondary Study Endpoints

The secondary study endpoint will be the potential efficacy of LLLT in HNC patients, including lymphedema progression, symptom burden, and functional status.

# 4 Study Population and Duration of Participation

### 4.1 Inclusion Criteria

- >18 years of age
- Completion of either postoperative radiation or chemoradiation therapy
- No evidence of cancer
- Having head and neck external lymphedema
- · Ability to speak and read English
- Able to provide informed consent

### 4.2 Exclusion Criteria

Patients will be excluded if they have any of the following medical conditions that would prohibit the safe implementation of LLLT: pregnancy; photosensitivity; chronic inflammatory diseases; venous thrombosis; history of severe trauma; medication that affects body fluid and electrolyte balance; use of high doses of non-steroidal anti-inflammatory drugs; or pre-existing skin rash, ulceration, open wound in the treatment area; and allergic and other systemic skin diseases. In addition, patients will be excluded if they are in active physical therapy and/or lymphedema therapy.

### 4.3 Subject Recruitment

The following recruitment procedures will be used: screening at HNC clinics and attendance at Head and Neck tumor board and case conferences. All direct patient recruitment activities will be conducted at the Penn HNC clinics where private rooms are available to be used for conducting clinical research projects.

### 4.4 Duration of Study Participation

The duration of the study subjects' participation will be 10 weeks, including screening, study intervention phase (6 weeks) and follow up time period (up to 4 weeks).

### 4.5 Total Number of Subjects and Sites

Total number of subjects: 25

Single-site study: Subjects will be enrolled at Penn only.

### 4.6 Vulnerable Populations

Not applicable.

### 5 Study Intervention (Study drug, device, biologic, vaccine, food etc.)

### 5.1 Description

The LTU-904 is a Class I laser device, which is a low output laser in the infrared wavelength (904nm) and no safety glasses are required as there is no risk of eye damage as defined by the standards set by the international Electrotechnical Commission.

### 5.2 Intervention Regimen

The LTU-904 will be used in the study. The following laser parameters commonly used in the literature will be used in the study: 5mW output; 904nm wavelength in pulsed mode; dosage (energy density) of 1.5J/cm<sup>2</sup>. For this pilot study, all the study participants will receive the same treatment regimen, including the same dose, therapy sessions, and treatment spots.

Participants will undergo the following procedures at each study visit. First, they will be asked to lie on a massage table. Then, the study lymphedema therapist will place a small laser device head directly on the skin of either left side or right side of the participant's face and neck, i.e., the side with the swelling and the tough/tight tissues. A total of 14 ~25 spots on the face and neck will be treated. The spots includes: maxillary prominence (1 spot), mandible (2 points), pre auricular (1 point), submental (3 points), sternocleidomastoid muscle (3 points), supraclavicular area (2 points), and scalene muscle (2 points). Each spot will be treated for about 60 seconds. Each study visit will take approximately 25-30 minutes. Prior to low-level laser therapy, participants will receive 5 minutes of simple manual lymphatic drainage (MLD) to the head and neck region that followed the international standards.

### 5.3 Storage

Study Device Storage, Delivery and Management: The LTU-904 will be purchased from RianCorp directly. The device will be shipped to the PI directly. The LTU-904 unit comes with a carry case that ensures the unit is stored safely. Both the PI Deng and the study lymphedema therapist (Joy Cohen) will be trained by an expert from RianCorp directly regarding how to store, dispense, and manage the device appropriately prior to subject enrollment or conducting research activity. The study lymphedema therapist will be responsible for storing, dispensing, and managing the laser device. The study lymphedema therapist will evaluate and monitor the LTU-904 unit regularly to ensure its normal function and prepare it for administration to subjects. The study lymphedema therapist will make sure the LTU-904 is stored properly after use of the device each time. The study lymphedema therapist will report the failed device to the PI Deng. The PI Deng will return the failed device to the manufacturer. The PI Deng will monitor the storage, delivery, and management of the laser device throughout the study.

### 5.4 Preparation and Packaging

The study lymphedema therapist (Joy Cohen) will properly prepare the LTU-904 unit for administration to subjects. Ms. Joy Cohen will make sure the LTU-904 is stored properly after use of the device each time.

### 5.5 Blinding

Not applicable.

### **Subject Compliance Monitoring** 5.6

The participants are encouraged to be compliant with the scheduled visits. The reasons for non-compliance with the study scheduled visits will be documented and potential underlying barriers will be explored.

### **Study Procedures and Data Collection**

### 6.1 Screening

The screening will be conducted by a trained staff member. Individuals who are interested in this research will be screened for eligibility for being in the study. A Screening Checklist will be used to ensure that eligible participants are enrolled in the study. A Recruitment Log will be used during the recruitment.

### 6.2 Study Intervention Phase

### 6.2.1 Visit 1: Baseline Visit

The following procedures and data collection will take place at study visit 1.

- Demographic Form
- Physical Exam for completing HN-LEF Grading Criteria
- Digital photographs of face and neck
- Modified Patterson Scale
- Symptom burden assessments (LSIDS-H&N and NDI)
- Functional status (neck range of motion)

In addition, the following variables will be abstracted from the medical chart with participants' permission.

- HNC Disease and treatment information (HNC Clinical Form)
- Lymphedema and fibrosis diagnosis and treatment information (LEF Treatment Form)

### 6.2.2 Visit 2: End of Intervention

The following procedures and data collection will take place at study visit 2.

- Physical Exam for completing HN-LEF Grading Criteria
- Digital photographs of face and neck
- Modified Patterson Scale
- Symptom burden assessments (LSIDS-H&N and NDI)
- Functional status (neck range of motion)

### 6.2.3 Visit 3: 4 – Week post Intervention

The following procedures and data collection will take place at study visit 3.

- Physical Exam for completing HN-LEF Grading Criteria
- Digital photographs of face and neck
- Modified Patterson Scale
- Symptom burden assessments (LSIDS-H&N and NDI)
- Functional status (neck range of motion)

### 6.3 Subject Withdrawal

Subjects may withdraw from the study at any time without impact to their care. They may be discontinued from the study at the discretion of PI Deng, due to lost follow-up or adverse events. Subjects may also be withdrawn by PI Deng from the study given safety consideration.

### 7 Statistical Plan and Statistical Analysis

While this study is a preliminary study of efficacy and effect sizes, a maximum alpha level of 0.05 will be used for the statistical tests.

Statistical analysis for primary aim (feasibility of the intervention): Descriptive statistical and graphical methods will summarize the rates of participation (recruited vs. consented), log data (e.g., sessions completed), completion of assessments throughout the study, adverse events (safety) and satisfaction data within both groups. It is expected that  $\geq 80\%$  of participants will complete the study activities, and  $\geq 80\%$  will report acceptable levels of satisfaction with the interventions, thereby demonstrating feasibility of the interventions proposed in this research.

For the secondary objective, change from baseline value will be computed for each outcome variable at each follow-up timepoint. The analysis of changes over time relies on mixed-effects modeling, which accounts for correlation among subjects' repeated measures using a compound symmetry covariance matrix. Results will be reported as model-based mean change ± standard error.

### 8 Safety and Adverse Events

### 8.1 Safety Monitoring

The following strategies will be in place to monitor safety of participants during the course of the study.

During the course of this study, study staff will observe for any adverse side effects or events when interacting with participants and be trained to report these to the PI's immediately. Common Terminology Criteria for Adverse Events (CTCAE version 4.03) will be used to document adverse events of the trial. All the staff members who are involved in this study will be trained how to use CTCAE version 4.03.

In addition, participants in this study will be screened against the inclusion and exclusion criteria. Participants will be educated regarding signs and symptoms related to adverse events (e.g., sudden increase in swelling) requiring urgent or emergent medical care.

### 8.2 Recording of Adverse Events

Each contact with the subject, the trained staff will seek information on adverse events by specific questioning and, as appropriate, by examination. Information on all adverse events will be recorded immediately in the source document, and also in the appropriate adverse event module of the case report form (CRF). All clearly related signs, symptoms, and abnormal diagnostic procedures results should recorded in the source document.

All adverse events occurring during the study period will be recorded. The clinical course of each event will be followed until resolution, stabilization, or until it has been determined that the study intervention or participation is not the cause. Serious adverse events that are still ongoing at the end of the study period will be followed up to determine the final outcome. Any serious adverse event that occurs after the study period and is considered to be possibly related to the study intervention or study participation will be recorded and reported immediately.

All adverse events will be reviewed by Drs. Deng and Lin, any contributing factors will be reviewed, and strategies to prevent further complications will be developed and implemented. Dr. Deng will meet with study staff monthly to evaluate any other safety concerns. Adverse events will be reported to the Penn IRB within the window required by the IRB. If study staff identify the following unanticipated problems related to the research (e.g., infection in the treated area, sudden increase in swelling), which occur during the study, Drs. Deng, Lin, and study lymphedema therapists will be notified immediately. Patients will be referred and received appropriate and timely therapy. Drs. Deng and Lin will determine if participants with adverse events or any unexpected issues will remain on the study based on safety consideration. Drs. Deng and Lin as well as the study lymphedema therapist will evaluate the relationship of each adverse event to the study procedures. PI Deng and Co-I Lin will be responsible for making the determination of the relationship

of the adverse event to the study procedures (e.g., definitely related, probably related, possible related, unlikely or unrelated).

# 8.3 Reporting of Adverse Events, Adverse Device Effects and Unanticipated Problems to Penn IRB and ACC

PI Deng and the study team will conform to the adverse event reporting timelines and formats, per the Penn IRB reporting requirements and Abramson Cancer Center reporting guidelines.

The following information will be included at the time of the initial report:

- Study identifier
- Study site
- Subject number
- A description of the event
- Date of onset

- Current status
- Whether study intervention was discontinued
- The reason why the event is classified as adverse events
- Investigator assessment of the association between the event and study intervention

Additionally all other events (unanticipated problems, adverse reactions, unanticipated adverse device effects and subject complaints) will be recorded and reported with respect to Penn policies as described in the Penn Manual.

### 8.3.1 Investigator reporting: notifying the study sponsor

Not applicable. The study has no external sponsor.

### 8.4 Stopping Rules

We do not anticipate significant adverse events. Given no safety data available in the population under study, the research may involve risks that are currently unforeseeable. If any one event is identified that may have caused any type of harm to a participant, study recruitment and associated study activities will be immediately halted until the study team reviews the event and determines if any study procedures need to be revised. Study recruitment and associated study activities will only resume after review of study protocol has been completed and any recommended revisions made as advised by both the study team and the Penn IRB.

### 8.5 Medical Monitoring

PI Deng will be responsible for overseeing the safety of the study. In addition, Co-I Lin (study physician) and Ms. Joy Cohen (study lymphedema therapist) will be involved in medical monitoring.

### 8.5.1 Data and Safety Monitoring Plan

The data and safety monitoring plan will adhere to policy guidance and standards set by the Penn IRB. The PI Deng will be responsible for monitoring the entire study.

Data Management: 1) Self-reported questionnaires will be completed by participants using a tablet to enter their responses into REDCap. The research assistant will review participants' completeness for each questionnaire. If participants prefer or if there are technical difficulties, hard copy forms will be used. All hard copy data will be double-entered into REDCap, checked for discrepancies, and reconciled with hard copy forms. All forms will be stored in a secured cabinet. 2) Phyiscal examination data collected by the study staff will be entered by the research assistant into REDCap. These data will also be double-entered, checked for discrepancies, and reconciled with the hard copy form. 3) Imaging data (digital photos) will be deidentified (white out eyes) and only scoring data will transfer out to REDCap. Data from various sources will be integrated into the study databases by the Data Specialist. All data will be coded without any identifiable information. The PI Deng and the data specialist will monitor and ensure that all data are timely entered into

the databases and all protocol specifics are met. PI Deng will monitor all databases monthly and maintain a master table that links participants to ID number in a password-protected database on a secure server throughout the study and after close of study.

Monitoring by the PI: PI Deng, with assistance from the Co-I Lin, the study lymphedema therapist (Joy Cohen), and other study staff members, will monitor all the study activities to ensure safety of participants and integrity of the data collection and management. The research team will meet monthly to discuss recruitment, retention, study progress, and any safety concerns. Any potential issues related to the study activities will be discussed and addressed appropriately and timely. Participants will be educated regarding signs and symptoms related to adverse events requiring urgent or emergent medical care. All adverse events will be documented using CTCAE criteria, reviewed by Drs. Deng and Lin. Any contributing factors will be reviewed. Strategies to prevent further complications will be developed and implemented. Although adverse events are highly unlikely, should they develop, they will be reported to the Penn IRB, within the required time window.

### 9 Study Administration, Data Handling and Record Keeping

# 9.1 Confidentiality

All the study data will be stored in a secured network drive managed by University of Pennsylvania School of Nursing IT staff member. All participants will be assigned a study ID number (e.g., 100). Numbers will be assigned by trained study staff. It is important and necessary for the study team to know participants names in order to communicate with them during the study. This information will be maintained in a participant tracking database that is not stored on the hard drive, accessible only to the study team members through a password protected computer and link to a Penn School of Nursing server that is accessible only the study team. The name column will be deleted at the end of the study.

### 9.2 Data Collection and Management

Data collection will be conducted by a trained staff member at a private room at the Abramson Cancer Center (ACC) HNC clinics (participant recruitment and baseline data collection). The following procedure will be utilized to protect the privacy of the research participant. All data will be coded and filed without any name or other identifiable information. Self-reported questionnaires will be completed by participants using an encrypted and secured tablet to enter their responses into REDCap. The research assistant will review participants' completeness for each questionnaire. If participants prefer or if there are technical difficulties, hard copy forms will be used. All hard copy data will be double-entered into REDCap, checked for discrepancies, and reconciled with hard copy forms. All hard copies will be placed in a locking file cabinet. Only the study team have access to the file cabinet and electronic database. After the study is concluded, the research data will be stored at Penn School of Nursing.

### 10 Study Monitoring, Auditing, and Inspecting

### 10.1 Study Monitoring Plan

Monitoring by the PI: The PI Deng, with assistance from the Co-I Lin, the study lymphedema therapist (Joy Cohen), and other study staff members, will monitor all the study activities to ensure safety of participants and integrity of the data collection and management. The research team will meet monthly to discuss recruitment, retention, study progress, and any safety concerns. Any potential issues related to the study activities will be discussed and addressed appropriately and timely. Participants will be educated regarding signs and symptoms related to adverse events requiring urgent or emergent medical care. All adverse events will be documented using CTCAE criteria, reviewed by Drs. Deng and Lin. Any contributing factors will be reviewed. Strategies to prevent further complications will be developed and implemented. Although adverse events are highly unlikely, should they develop, they will be reported to the Penn IRB, within the required time window.

### 10.2 Auditing and Inspecting

The PI Deng will permit study-related monitoring, audits, and inspections by the IRB, government regulatory bodies, and University compliance and quality assurance groups of all study related documents (e.g., source documents, regulatory documents, data collection instruments, study data etc.).

### 11 Ethical Considerations

Although this is an interventional study, foreseeable physical, psychological, financial, legal, or other risks from study participation are believed to be minimal.

### 11.1 Risks

- 1) Physical: No physical risks (e.g., worsening lymphedema or fibrosis) from using LLLT in individuals with breast cancer-related lymphedema have been reported in the known current literature review. No physical risks from using LLLT were reported in the cases studies conducted in individuals with head and neck lymphedema. Subjects will not have any burning sensation, warmth, or any other uncomfortable sensations on the sites treated with low-level laser. Currently, there is no safety data in the population under study. Thus, we will inform participants of reporting any physical damages they have during the course of the study.
- 2) Psychological: There are no known psychological risks associated with LLLT.
- 3) Financial: The LLLT will be provided free of charge. Patients may incur expense of gas when driving to the Penn Clinic.
- 4) Legal: There are no known legal risks.
- 5) Other: There may be risks that are unknown at this time.

Our planned protections from the above-noted risks are as follows:

- 1) Physical: Currently, there are no known potential physical risks for being in this study. Given no safety data available in the population under study, the research may involve risks that are currently unforeseeable. To minimize any potential physical risks, the following will be done: a) Participants will be given the study contact phone numbers and emails to ask any questions or to report any unexpected problems if the problems are directly related to the study activities; b) if study staff identify any unanticipated problems, Drs. Deng, Lin, and study lymphedema therapist (Joy Cohen) will be notified immediately. Appropriate evaluation and timely therapy will be provided to the participant. Deng, Lin, and study lymphedema therapists will determine if participants with significant unanticipated issues will remain on the study based on safety consideration; and c) if anyone experience an adverse event directly related to the study activities that are done for research, they can get reasonable, immediate, and necessary medical care for their adverse events at Penn.
- 2) Psychological: If study staff identifies participants with significant distress during the course of the study, PI Deng and Co-I Lin will be notified immediately so that appropriate psychological evaluation and referrals will be made. Drs. Deng and Lin will determine if participants with significant psychological issues will remain on study.
- 3) Financial: The LLLT will be provided free of charge. Patients will incur expense of gas when driving to the Penn Clinic during study follow-up visits. To offset travel/gas cost, participants will be provided a financial token of appreciation for participation in the study.
- 4) Legal: There are no known legal risks.
- 5) Other: Should the team become aware of any additional risks, participants will be notified and informed consents will be modified to reflect the new information.

# 11.2 Benefits

Potential benefits to the individual: Although the potential direct benefit to study participants is unknown, individual participants will be exposed to and have increased knowledge about lymphedema and fibrosis. Participants may have positive feelings about participation in a research program that may benefit others.

Potential benefits to human kind: Possible future benefits for HNC survivors are potentially substantial. If we are able to demonstrate that LLLT is safe, feasible and effective in HNC patients, we will be adding to the armamentarium of an alternative intervention that can diminish progression of lymphedema and fibrosis, decrease symptom burden, increase function, and improve overall quality of life.

### 11.3 Risk Benefit Assessment

Currently, there are no known potential risks for being in this study. Given no safety data available in the population under study, the research may involve risks that are currently unforeseeable. As noted above, potential benefits are reasonable and substantial. Thus, based on the risk benefit assessment, it appears to be acceptable for this research within human subjects.

### 11.4 Informed Consent Process / HIPAA Authorization

Once the study is approved by the Penn IRB and the ACC, the trained study team members will meet with potential participants who express interest in the study. Potential study participants will be provided one copy of the informed consent to read and review. Study team members will review the study procedures and activities with potential participants. The informed consent document will be written in lay language and cover all study activities participants will engage in during the study, define the length of time the study will be conducted, and provide instructions for participant withdrawal from the study should they choose to do so. Study staff will review and, when necessary, read the informed consent document to potential participants. Participants will be given ample time and opportunity to ask questions, and all questions will be answered by study staff. The consent process will take place in a private location, with a closed door. Once participants have had an opportunity to ask questions, those questions have been answered, and they indicate an interest in participation, they will be asked to sign a written informed consent document as the study staff witnesses. In addition, the participant will be given a copy of informed consent signed by both the participant and study staff. We will not seek waivers of the informed consent process.

### 12 Study Finances

# 12.1 Funding Source

Not applicable.

# 12.2 Conflict of Interest

All the team members will follow the University of Pennsylvania Policy on Conflicts of Interest Related to Research.

### 12.3 Subject Payments

All participants will be provided with a financial token of appreciation that increases slightly the longer they are in the study (\$15 for baseline, \$20 for end of intervention, \$20 for 4-week post-intervention, and \$25 for 8-week post-intervention).

### 13 Benchmarks for Study/Publication Plan

The key benchmark for success of this study is to complete recruitment goals and data collection as scheduled. The information gathered from this study will provide important data for designing a large clinical trial that tests the efficacy of LLLT on lymphedema in the HNC survivors. Additional benchmarks for success include: 1) dissemination of preliminary findings at professional conferences and 2) submission of articles to peer-reviewed journals.